CLINICAL TRIAL: NCT05037136
Title: Remote Monitoring of AF Recurrence Using mHealth Technology (REMOTE-AF)
Brief Title: Remote Monitoring of AF Recurrence Using mHealth Technology
Acronym: REMOTE-AF
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 283058
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Long Standing Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Digital health; Artificial intelligence; Catheter ablation; Thoracoscopic surgical AF ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ablation: Participants recruited from the LoTO_CASA_AF trial (ClinicalTrials.gov Identifier: NCT04280042) who underwent either conventional catheter ablation or thoracoscopic surgical ablation to treat their long standing persistent AF with be asked to continue downloading data from their implanted loop recorder and monitor their heart rate and physical activity level (step count) using a wrist worn activity tracker.

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia worldwide. It carries a significant health burden, conferring on sufferers a reduction in quality of life, risk of significant morbidities such as stroke and heart failure, and significant mortality. At present, diagnosis of AF involves referral for conventional 12 lead electrocardiogram (ECG) recording, ambulatory ECG for fixed time period recording, or insertion of implantable loop recorders (ILR). These investigations are limited both by recording only at specific time points and failing to explore the interaction between heart rate and day-to-day physical activity. In recent years, the use of mobile health (mHealth) devices has emerged as a direct-to-consumer option for monitoring parameters such as heart rate and activity levels. From a clinical perspective they potentially offer a less invasive and cost-effective investigative approach, with remote monitoring solution to identify and possibly predict AF. In this study, the investigators propose to recruit participants who have undergone an ablative procedure as part of a randomised clinical trial (LoTO in CASA LSPAF: NCT04280042) and monitor for recurrence of AF using mHealth technology by correlating with ILR data.

ELIGIBILITY:
Inclusion Criteria:

* Participants in LoTO in CASA LSPAF with implanted loop recorders (ILR)

Exclusion Criteria:

* Participants in LoTO in CASA LSPAF who had their ILR explanted

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with long standing persistent atrial fibrillation who have undergone an ablative procedure for the condition and who were implanted with a loop recorder to monitor their heart rhythm as part of their participation in LoTO in CASA LSPAF (NCT04280042)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
To explore if mHealth obtained heart rate (PPG) data can be correlated to recurrence of AF/AT in patients who have undergone an ablative procedure. | 18 months
  Exploring a correlation between PPG data from a wrist worn device and atrial arrhythmias recorded by implantable loop recorder or other clinically indicated rhythm recording device.

CONTACTS AND LOCATIONS:
Overall Officials: Shouvik Haldar, Principal Investigator — Royal Brompton & Harefield Hospitals, GSTT NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield Hospitals, GSTT NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adasuriya G, Barsky A, Kralj-Hans I, Mohan S, Gill S, Chen Z, Jarman J, Jones D, Valli H, Gkoutos GV, Markides V, Hussain W, Wong T, Kotecha D, Haldar S. Remote monitoring of atrial fibrillation recurrence using mHealth technology (REMOTE-AF). Eur Heart J Digit Health. 2024 Feb 12;5(3):344-355. doi: 10.1093/ehjdh/ztae011. eCollection 2024 May. PMID 38774381